CLINICAL TRIAL: NCT05963308
Title: Promoting Sustainable Return to Work Among Employees on Sick Leave Due to a Mental Health Condition: Evaluation of the HealthyMinds Online Group Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université du Québec a Montréal (Other)
Collaborators: Ciusss de L'Est de l'Île de Montréal (Other); PhysioExtra (Unknown); Energir (Unknown)
Responsible Party: Principal Investigator, Marc Corbière, Full Professor, Université du Québec a Montréal
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2023-0SYA-316461
Record Dates: First submitted 2023-07-18; First posted 2023-07-27 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Depression Anxiety Disorder; Adjustment Disorders; Adjustment Disorder With Anxious Mood; Adjustment Disorder With Depressed Mood
MeSH Terms: conditions — Adjustment Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online group intervention "Healthy Minds" (Experimental)
  Interventions: Behavioral: Healthy Minds
- Control group (No Intervention): Like the intervention group, the control group will complete an online set of questionnaires at the following time points:
  * Baseline
  * First follow-up (2 months after baseline)
  * Second follow-up (6 months after baseline)
  * Third follow-up (12 months after baseline)
  The questionnaires will cover the following domains:
  * Sociodemographic and biopsychosocial factors
  * Symptoms associated with the primary mood disorder
  * Cognitive difficulties and distortions
  * Self-efficacy in relation to returning to work
  * Work accommodations and natural supports
  * Relationship with immediate supervisor
  * Work functioning
  * Return-to-work time (number of days away from work)

INTERVENTIONS:
Behavioral: Healthy Minds — The group intervention (approximately 5 participants per group, 8 groups) is facilitated by two clinicians and consists of 8 sessions (one per week for 8 weeks), with each session focusing on a specific aspect of the return-to-work process from a cognitive-behavioral perspective:
  Week1: Coping with work stress at work W2 and W3: Recognizing and modifying my dysfunctional beliefs linked to work W4: Overcoming obstacles linked to work functioning and maintaining work W5: To put in place needed work accommodations with the support of the immediate supervisor W6: My strengths and competencies related to work W7: Accepting criticism and asserting myself appropriately W7: My strengths and related skills W8: My best coping strategies for work Both intervention and control participants receive their standard individualized care from their clinician. However, for the experimental participants, the Healthy Minds intervention is an added component to their regular care.
  Arms: Online group intervention "Healthy Minds"

SUMMARY:
The purpose of this clinical trial is to evaluate the impact of an online group intervention called Healthy Minds in facilitating a sustainable return to work for individuals with a mood disorder. The study aims to answer the following key questions :

* Does receiving the Healthy Minds online intervention lead to a more sustainable return to work compared to not receiving the intervention?
* Are the health outcomes (e.g., depressive symptoms) and work-related outcomes (e.g., work functioning) of individuals who receive the Healthy Minds online intervention better than those who do not receive the intervention in the year following the intervention?

Both experimental and control participants will be recruited at baseline while on sick leave (expected to return to work in less than one month) or recently returned to work (less than one month). Participants will complete a series of online questionnaires at the following time points :

* Baseline
* First follow-up (2 months after baseline)
* Second follow-up (6 months after baseline)
* Third follow-up (12 months after baseline)

The questionnaires will cover the following areas :

* Sociodemographic and biopsychosocial factors
* Symptoms associated with the primary mood disorder
* Cognitive difficulties and biaises
* Self-efficacy related to return to work
* Work accommodations and natural supports
* Relationship with immediate supervisor
* Work functioning
* Return to work time (number of days away from work)

Experimental participants will participate in the 2-month online Healthy Minds group intervention (cohort of 5 participants) between the baseline assessment and the first follow-up. The intervention consists of 8 sessions (one per week for 8 weeks), with each session focusing on a specific aspect of the return-to-work process from a cognitive-behavioral perspective.

ELIGIBILITY:
Inclusion Criteria:

* Be in the process of returning to work after depression, anxiety disorder, adjustment disorder (with depressed mood, or anxious mood).

or

* Been back for less than a month

Exclusion Criteria:

* Inability to communicate in French
* Have a known organic disorder
* Have already received CBT-type intervention (group or individual)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-03-06 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Sustainable return-to-work | Baseline; follow-ups at six months and 12 months
  The number of days of job retention after returning to work
Depressive symptoms | Baseline; follow-ups at two months, six months and 12 months
  Patient Health Questionnaire for depression (PHQ-9)
Anxiety symptoms | Baseline ; follow-ups at two months, six months and 12 months
  Generalized Anxiety Disorder Scale (GAD-7)
Work functioning | Follow-ups at six months and 12 months
  Endicott Work Productivity Scale (EWPS)
Relationship with immediate supervisor | Follow-ups at six months and 12 months
  Inventory of perceptions of supervisory style at work
Work accommodations | Follow-ups at six months and 12 months
  The Work Accommodation and Natural Support Scale (WANSS).
Return to Work Obstacles and Self-Efficacy | Baseline ; Follow-ups at two months
  Return to Work Obstacles and Self-Efficacy Scale (ROSES)
Cognitive difficulties | Baseline ; Follow-ups at two months, six months and 12 months
  Online Stroop test (French version)
Cognitive biases | Baseline ; Follow-ups at two months, six months and 12 months
  Davos Assessment of the Cognitive Biases Scale

CONTACTS AND LOCATIONS:
Overall Officials: Marc Corbière, PhD, Principal Investigator — Université du Québec a Montréal
Locations (1):
- Université du Québec à Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No